CLINICAL TRIAL: NCT04165746
Title: Early Institutionalization Intervention Impact Project
Acronym: EI-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Maryland, College Park (Other); Tulane University (Other); Instituto PENSI (Unknown); Harvard University (Other); Inter-American Development Bank (Other); Lumos Foundation (Unknown); Two Lilies Fund (Unknown); Fundaçao Maria Cecilia Souto Vidigal (Unknown)
Responsible Party: Principal Investigator, Charles Alexander Nelson III, Richard David Scott Chair in Pediatric Developmental Medicine Research, Professor of Pediatrics and Neuroscience, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-P00026292
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-05

CONDITIONS: Socioemotional Development; Cognitive Ability; Behavioral and Neural Patterns of Attention; Brain Function; Psychopathology
Keywords: Brazil; children; foster care; institutionalization; attachment; brain function; language; growth; Intelligence Quotient (IQ); early intervention
MeSH Terms: conditions — Behavior; Language | interventions — Foster Home Care

STUDY DESIGN:
Intervention Model Description: Children will be randomized to either enhanced institutional care or enhanced foster care. Both arms of the RCT will participate in an intervention. Children randomized to foster care will receive 2 forms of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Institutional Care (Experimental): Caregivers at institutions will participate in a caregiving training, called Attachment VideoFeedback Intervention (AVI). During AVI a trained interventionist meets with a caregiver and child in the home environment.
  The AVI Interventionist will meet with caregivers and children for 8, 1.5-hours sessions over 8-9 weeks to discuss recordings of children and their caregivers. As described above, the sessions will focus on creating a positive atmosphere by reinforcing positive interactions.
  Interventions: Behavioral: Caregiving Intervention
- Enhanced Foster Care (Experimental): Foster parents will be recruited, consented to background checks, and trained in Portuguese. Hired foster parents will supported and monitored by project social workers and psychologists from local Foster Care programs. Foster parents will received frequent visits from the social workers, with visits occurring weekly for several months after placement of the child, then biweekly and later monthly. Project social workers will consult weekly with US staff experienced in dealing with young children in foster care.
  Additionally, foster parents will participate in the VIPP caregiving training, in the same format as that described in the Enhanced Institutional Care Arm: the VIPP Interventionist will meet with caregivers and children for 5, 2-hours sessions over 6-8 weeks to discuss recordings of children and their caregivers. As described above, the sessions will focus on creating a positive atmosphere by reinforcing positive interactions.
  Interventions: Other: Foster Care; Behavioral: Caregiving Intervention

INTERVENTIONS:
Other: Foster Care — Upon entry into the Child Protection System, if the child is assigned to one of the districts participating in the RCT, the court will notify the study team. Children that have been randomly assigned to Foster Care will be placed in a foster home within 48 hours of referral to the Family Court/Child Protection System.
  Children and Foster Parents will receive biweekly visits from Social Workers. Children and Foster parents will also participate in the caregiving intervention described below. Children will remain in the placement until such time as the social workers, psychologists and Family Court Judge determine that one of the following outcomes is appropriate: reunification with biological family or adoption.
  Arms: Enhanced Foster Care
Behavioral: Caregiving Intervention — During AVI an intervenor meets with a caregiver (foster parent or caregiver at the institution) and child in the home environment. During each session, the intervenor videotapes the caregiver and child doing play-based activities. During that meeting, the intervenor reviews the videos with the caregiver and provides positive, constructive feedback to the caregiver. AVI is aimed at increasing sensitivity in parents/caregivers in order to encourage positive interactions. The guiding principles are to create a positive environment and to convey that the caregiver is the expert on their own child. The AVI methodology was selected to be used as a method of caregiving intervention with the study participants due to its demonstrated results in its use with children in contexts of social vulnerability, as well as families included in the child protection system. This will be the first time that AVI is being used in foster and institutional care in Brazil.
  Other Names: Attachment Video Feedback intervention

SUMMARY:
The purpose of this study is to determine the effects of early intervention (placement into foster care, and a caregiving training) on physical, cognitive, social and brain development and psychiatric symptomatology in children place in out-of-home care.

DETAILED DESCRIPTION:
The Early Institutionalization Intervention Impact (EI-3) Project will document and compare the impact of enhanced institutional care on early childhood development to that of high-quality foster care. We will recruit a large (n= 220) samples of young children who have been identified as having to be removed from their families and we will randomize these children to two groups: enhanced institutional care (Group 1) or to enhanced foster care (Group 2). Institutional caregivers and Foster Parents will participate in a caregiving training, along with the child, that includes 8-1.5 hour sessions over 8-9 weeks.

In this Randomized Control Trial (RCT), we will assess the children in Groups 1 and 2 at the time they come into care and then at several follow-up time points (12 months, 24 months, 36 months of age). We hypothesize that children placed into foster/family care (FCG) will display enhanced socioemotional development, and enhanced behavioral and neural patterns of attention, cognition and social cognition, compared to children placed in enhanced institutional care.

ELIGIBILITY:
Inclusion Criteria:

* newly entering the institution system in and near São Paulo, Brazil, and the institution director or foster parent is the guardian at the time of baseline,
* at the time of baseline assessment the child is less than 24 months old,
* the child's birth weight must be at or above 2500 grams; none should be small or large for dates.

Exclusion Criteria:

* the child does not have a neurological or other genetic condition that severely impairs typical development (e.g. Cerebral Palsy, Fetal Alcohol Syndrome, Down Syndrome)
* the child is below 2500 grams.

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Differences in security of attachment | baseline, 12 mos, 24 mos, 36 mos
  Strange Situation Procedure
Differences in Alpha Electroencephalogram (EEG) Power, Coherence and Functional Connectivity | baseline, 12 mos, 24 mos, 36 mos
  EEG power

SECONDARY OUTCOMES:
Differences in Cognition in early Childhood | baseline, 12 mos, 24 mos, 36 mos
  Mullen Scales of Early Learning, AGS Edition. For the subscales (Visual Receptions, Fine Motor, Gross Motor, Receptive, and Expressive Language), the minimum T-score is 20 and the maximum is 80. A higher score indicates a better outcome. The Composite Standard Score goes from 49 to 155; 155 is the best outcome.
Differences in Attachment Disturbances and Disorders | baseline, 12 mos, 24 mos, 36 mos
  Disturbances of Attachment Interview
Differences in Competence | baseline, 12 mos, 24 mos, 36 mos
  Infant Toddler Social Emotional Assessments- Revised. Range for competence is 0-66. Ratings are 0, 1, 2 on 33 items. Higher scores are better outcomes. T-scores of 35 or lower on the Competence scale are also termed "of concern."

CONTACTS AND LOCATIONS:
Overall Officials: Nathan A Fox, PhD, Principal Investigator — University of Maryland; Charles A Nelson, PhD, Principal Investigator — BOSTON CHILDRENS HOSPITAL/ Harvard University; Charles H Zeanah, PhD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Instituto PENSI, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No